CLINICAL TRIAL: NCT03415581
Title: Doxazosin: Evaluation of Its Ability to Alter the Abuse Liability of Oxycodone in Humans
Brief Title: Evaluation of Doxazosin to Alter the Abuse of Oxycodone
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated by sponsor due to bad risk/benefit ratio.
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Sandra D. Comer, Research Scientist/Professor of Clinical Neurobiology (In Psychiatry), New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 7547
Record Dates: First submitted 2018-01-11; First posted 2018-01-30 (Actual); Results first posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-03

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Doxazosin (Placebo First) (Placebo Comparator): Maintenance on a daily dose of oral doxazosin (0 mg) for 4 weeks, followed by 4-week maintenance on active doxasozin (up to 16mg/day or the highest tolerated dose. During this time subjects complete testing sessions (Self-administration, Cue session) assessing the abuse potential of intranasal oxycodone.
  Interventions: Drug: Intranasal Oxycodone; Behavioral: Cue Session
- Doxazosin (Active First) (Active Comparator): Maintenance on a daily dose of oral doxazosin (16 mg, or the highest tolerated dose) for 4-weeks, followed by 4-week maintenance on placebo doxasozin. During this time subjects complete testing sessions (Self-administration, Cue session) assessing the abuse potential of intranasal oxycodone.
  Interventions: Drug: Intranasal Oxycodone; Behavioral: Cue Session

INTERVENTIONS:
Drug: Intranasal Oxycodone — Under each doxazosin maintenance condition the effects of intranasal oxycodone will be assessed in order to determine if doxazosin reduces dependent measures assessing its abuse potential.
  Other Names: Oxycodone HCl
Behavioral: Cue Session — During the cue exposure session participants are presented with neutral cues followed by drug-related cues. This procedure will allow the investigators to determine whether the study medication affects reactivity to drug-related cues.

SUMMARY:
Healthy, adult men and women, aged 21 to 59 years, who abuse opioids and are physically dependent on them will be recruited to participate in a study to examine the ability of doxazosin, an epinephrine receptor blocker, to alter the abuse potential of oxycodone. After participants complete the screening process, they will be scheduled for inpatient admission onto our clinical inpatient where they will reside during the 8-week study. During Weeks 1-2, participants will be transitioned from their normal opioid use regime onto oral morphine until withdrawal dissipates. At this time participants will also be stabilized on the first dose of doxazosin (0 or 16 mg/day; active doxazosin will be started at 4 mg and increased by 4 mg every 3 days). During Weeks 3-4, either active or placebo oxycodone will be available (in random order). Monday-Friday each these drugs will be tested using our sample and choice self-administration procedure. On Friday, participants will also complete a cue exposure session during which they will be presented drug cues to determine whether the study medication affects how participants react to them. To summarize, Weeks 1-2 and 5-6 will be stabilization weeks (0 or 16 mg doses of doxazosin administered in random order) and Weeks 3-4 and 7-8 will be test weeks under each of the doxazosin maintenance doses. At the conclusion of the study, participants will be given an exit interview, warnings about re-initiation of opioid use, and counseling about the different treatment options for Opioid Use Disorder. Within 1 week after discharge, investigators will assess adverse events using the a number of clinical assessments. At each weekly visits, investigators will assess participants' interest in treatment and drug use patterns.

DETAILED DESCRIPTION:
Healthy, adult men and women, aged 21 to 59 years, who abuse opioids and are physically dependent on them will be recruited to participate in a study to examine the ability of doxazosin, an alpha-1 adrenergic receptor antagonist, to alter the abuse liability of oxycodone. After participants complete the screening process, they will be scheduled for admission onto the General Clinical Research Unit on 5-South where they will reside during an 8-week study . During Weeks 1-2, participants will be stabilized on morphine and the first dose of doxazosin (0 or 16 mg/day; active doxazosin will be started at 4 mg and increased by 4 mg every 3 days; dosing will occur at 8pm each evening). During the stabilization periods, participants will be treated for emergent withdrawal symptoms with supplemental medications until withdrawal symptoms have dissipated.

During Weeks 3-4, either active or placebo oxycodone will be available (order of testing active or placebo oxycodone will be randomized). During active oxycodone weeks, participants will receive a sample dose of intransasal (IN) oxycodone (0, 12.5, 25, 50, or 100 mg/70kg) during morning sessions on Monday-Friday. The sampled reinforcer will be available during afternoon choice sessions using a modified progressive ratio self-administration procedure. During placebo oxycodone weeks, participants will receive a sample dose of placebo oxycodone (0 mg/70kg) during morning sessions on Monday-Thursday followed by afternoon choice sessions. On Friday, participants will receive 25 mg IN oxycodone during a sample session (the oxycodone dose on Fri morning will always be active). When self-administering oxycodone, participants will be instructed to insufflate the entire dose through one or both nostrils within 5-10 seconds. Following the sample session on Fri, participants will complete a cue exposure session during which they will be presented with neutral cues followed by drug cues. This procedure will allow the investigators to determine whether the study medication affects reactivity to drug-related cues after a period of no oxycodone availability. After the cue exposure session on Fri, participants will be given the opportunity to self-administer oxycodone. To summarize, Weeks 1-2 and 5-6 will be stabilization weeks (0 or 16 mg doses of doxazosin administered in random order) and Weeks 3-4 and 7-8 will be test weeks under each of the doxazosin maintenance doses. At the conclusion of the study, participants will be given an exit interview during which the study will be described. Those who are interested in treatment for their drug use at the end of the study will be offered referrals to studies at our Substance Treatment and Research Service or other treatment providers. Within 1 week after discharge, investigators will assess adverse events, pregnancy (using a urine pregnancy test), general health (complete blood count, blood chemistry, urinalysis, blood pressure, heart rate, body weight, EKG), and suicide (Columbia Suicide Severity Rating Scale).

ELIGIBILITY:
Participants must meet all of the following inclusion criteria to be enrolled into the study:

1. 21-59 years of age. Ascertained by: Self-reported age and/or verification with legal identification.
2. Diagnostic criteria for Opioid Use Disorder moderate-severe (304.00) as per DSM-V Ascertained by: Clinical interviews (telephone, psychologist, nurse, physician), naloxone challenge test/visual evidence of opioid withdrawal.
3. No current or past diagnosis of schizophrenia, schizoaffective disorder, or other psychotic disorder; bipolar I or bipolar II disorder, other major mood, psychotic, or anxiety disorder that might interfere with the study. Ascertained by: Clinical interview with physician or nurse.
4. Physically healthy. Ascertained by: Clinical interview with physician, laboratory tests (urinalysis, blood chemistry, 12-lead ECG), physical examination, self-reported medical history.
5. Able to perform study procedures. Ascertained by: Practice session or Clinical Judgement (Psychologist or Physician)
6. Normal body weight. Ascertained by: Body Mass Index <30.
7. Current or history of intranasal opioid use. Ascertained by: Clinical interviews (telephone, psychologist, and psychiatric NP, or physician).
8. Current intranasal or intravenous use of opioids in amounts and/or frequencies that meet or exceed those used in the proposed study (e.g., 3-4 tablets of a prescription opioid medication per day or 1-2 bags of heroin per day). Ascertained by: Clinical interviews (telephone, psychologist, psychiatric NP, or physician)
9. If female and using oral contraceptives, must use alternative forms of contraception as well (e.g. condoms in combination with spermicide). Ascertained by: Clinical interviews (telephone, psychologist, nurse, physician), physical examination.
10. Has not participated in another opioid laboratory study within the past 3 months. Ascertained by: Clinical interviews (psychologist physician, or psychiatric NP), review of laboratory records.

Participants will be excluded from study participation if they meet any of the following exclusion criteria:

1. Meeting DSM-V criteria for substance use disorder (moderate-severe) on drugs other than opioids, nicotine or caffeine (must be less than 500 mg caffeine daily). Ascertained by: Clinical interview with physician or psychiatric NP, urine screen, observation.
2. Participants requesting treatment. Ascertained by: Self-report during interview.
3. Treatment with any investigational drug during the last 30 days. Ascertained by: Self-report during interview.
4. Participants on parole or probation. Ascertained by: Self-report during interview, criminal background check upon admission.
5. Currently pregnant or trying to conceive, or currently lactating. Ascertained by: Blood pregnancy testing at screening, on admission and (beta hCG), and self-report during interview and study visits.
6. Current or recent history of significant violent or suicidal behavior and/or suicidal/homicidal risk. Ascertained by: Clinical interview with a psychiatrist or psychiatric NP, and C-SSRS, MINI, and Beck Depression Inventory (based on current state and history).
7. Cannot read or understand the self-report assessment forms unaided, or are so severely disabled that they cannot comply with the requirements of the study. Ascertained by: Clinical interview (psychologist, physician, or psychiatric NP), or practice session.
8. Elevated liver function tests (i.e., AST and ALT > 3 times the upper limit of normal (ULN); bilirubin > 2x ULN; hepatitis B or chronic hepatitis C). Ascertained by: Laboratory tests.
9. Physical disorders that might make participation hazardous such as AIDS, cancer, baseline hypotension, orthostatic hypotension or syncope, hypertension (blood pressure > 140/90), uncontrolled diabetes, pulmonary hypertension or heart disease (please note that participants will be asked about previous visits to a cardiologist, chest pain, or strong palpitations; if these exist, they will be referred to a cardiologist and excluded unless cleared for participation by a cardiologist). Ascertained by: Clinical interview (psychologist, physician, or psychiatric NP) physical examination, 12-lead ECG.
10. Current major Axis I psychopathology other than opioid use disorder (e.g., mood disorder with functional impairment or suicide risk, schizophrenia), that might interfere with ability to participate in the study. Ascertained by: Clinical interviews (psychologist, physician, or psychiatric NP).
11. Sensitivity, allergy, or contraindication to opioids, doxazosin, adrenergic antagonists or agonists, or similar compounds. Ascertained by: Clinical interview (psychologist, physician, or psychiatric NP).
12. Planning to conceive within 6 months of study participation. Ascertained by: Clinical interview (psychologist, physician, or psychiatric NP).
13. Use of any prescription, over-the-counter medication that affects CYP3A4 activity are prohibited for at least 7 days prior to the anticipated study start date; or the use of phosphodiesterase inhibitors and MAOIs 14 days prior to the study. Ascertained by: Medical History, Clinical Interview ((psychologist, physician, or psychiatric NP).

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2017-02-12 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra D Comer, PhD, Principal Investigator — NYSPI/CUMC
Locations (1):
- Jermaine Jones, Manhattan, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Doxazosin, Then Active Doxazosin: Maintenance on a daily dose of oral doxazosin (0 mg) for 4 weeks. During this time subjects complete testing sessions (Self-administration, Cue session) assessing the abuse potential of intranasal oxycodone.
  Intranasal Oxycodone: Under each doxazosin maintenance condition the effects of intranasal oxycodone will be assessed in order to determine if doxazosin reduces dependent measures assessing its abuse potential.
  Cue Session: During the cue exposure session participants are presented with neutral cues followed by drug-related cues. This procedure will allow the investigators to determine whether the study medication affects reactivity to drug-related cues.
- Active Doxazosin the Placebo Doxazosin: Maintenance on a daily dose of oral doxazosin (16 mg) for 4 weeks. During this time subjects complete testing sessions (Self-administration, Cue session) assessing the abuse potential of intranasal oxycodone.
  Intranasal Oxycodone: Under each doxazosin maintenance condition the effects of intranasal oxycodone will be assessed in order to determine if doxazosin reduces dependent measures assessing its abuse potential.
  Cue Session: During the cue exposure session participants are presented with neutral cues followed by drug-related cues. This procedure will allow the investigators to determine whether the study medication affects reactivity to drug-related cues.
Period: Overall Study
Arm/Group | Placebo Doxazosin, Then Active Doxazosin | Active Doxazosin the Placebo Doxazosin
Started (Enrollment numbers are shown as a function of participants who were randomized to placebo (N=7) and active doxazosin (N=6) first. Prior to testing under active and placebo conditions participants completed stabilization on each medication "Stabilization" (Weeks 1-2 and 5-6), prior to testing under each medication "Testing" (Weeks 3-4 and 7-8). Thus, for the entire duration of the trial was 8 weeks for each participant (who completed).) | 7 | 6
Completed | 1 | 1
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Doxazosin (Placebo First): Maintenance on a daily dose of oral doxazosin (0 mg) for 4 weeks followed by active maintenance on doxazasin 16 mg (or the highest tolerated dose) for 4 weeks. During this time subjects complete testing sessions (Self-administration, Cue session) assessing the abuse potential of intranasal oxycodone.
  Intranasal Oxycodone: Under each doxazosin maintenance condition the effects of intranasal oxycodone will be assessed in order to determine if doxazosin reduces dependent measures assessing its abuse potential.
  Cue Session: During the cue exposure session participants are presented with neutral cues followed by drug-related cues. This procedure will allow the investigators to determine whether the study medication affects reactivity to drug-related cues.
- Doxazosin (Active First): Maintenance on a daily dose of oral doxazosin (up to 16 mg, or the highest tolerated dose) for 4 weeks, followed by maintenance on doxazosin 0 mg for 4 weeks. During this time subjects complete testing sessions (Self-administration, Cue session) assessing the abuse potential of intranasal oxycodone.
  Intranasal Oxycodone: Under each doxazosin maintenance condition the effects of intranasal oxycodone will be assessed in order to determine if doxazosin reduces dependent measures assessing its abuse potential.
  Cue Session: During the cue exposure session participants are presented with neutral cues followed by drug-related cues. This procedure will allow the investigators to determine whether the study medication affects reactivity to drug-related cues.
- Total: Total of all reporting groups
Arm/Group | Doxazosin (Placebo First) | Doxazosin (Active First) | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (10.4) | 47.7 (9.3) | 47.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 3 | 2 | 5
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Opioid Self-administration
Description: Clinical laboratory task where the participant is asked to choose between drug and money. Shown as the mean percent of drug choices.
Time Frame: Averaged across the 8-week trial.
Population: The number of participants analyzed for the measure represents 2 individuals who completed testing under both doxazosin and placebo maintenance conditions.
Measure: Mean (Standard Deviation); unit: Mean percentage of Drug Choices
Groups:
- Placebo: Maintenance on a daily dose of oral doxazosin (0 mg) for 4 weeks. During this time subjects complete testing sessions (Self-administration, Cue session) assessing the abuse potential of intranasal oxycodone.
  Intranasal Oxycodone: Under each doxazosin maintenance condition the effects of intranasal oxycodone will be assessed in order to determine if doxazosin reduces dependent measures assessing its abuse potential.
  Cue Session: During the cue exposure session participants are presented with neutral cues followed by drug-related cues. This procedure will allow the investigators to determine whether the study medication affects reactivity to drug-related cues.
- Doxazosin: Maintenance on a daily dose of oral doxazosin (16 mg) for 4 weeks. During this time subjects complete testing sessions (Self-administration, Cue session) assessing the abuse potential of intranasal oxycodone.
  Intranasal Oxycodone: Under each doxazosin maintenance condition the effects of intranasal oxycodone will be assessed in order to determine if doxazosin reduces dependent measures assessing its abuse potential.
  Cue Session: During the cue exposure session participants are presented with neutral cues followed by drug-related cues. This procedure will allow the investigators to determine whether the study medication affects reactivity to drug-related cues.
Arm/Group | Placebo | Doxazosin
Number analyzed (Participants) | 2 | 2
Mean percentage of Drug Choices
  Oxycodone 50 mg | 45 (.26) | 46 (.03)
  Oxycodone 0 mg | 33 (.92) | 38 (.57)
  Oxycodone 12.5 mg | 40 (.44) | 47 (.16)
  Oxycodone 100 mg | 46 (.03) | 44 (.21)
  Oxycodone 25 mg | 43 (.07) | 44 (.04)

2. Secondary Outcome: Opioid Craving
Description: Self-reported craving for opioid drugs. Participants are asked to indicate the extent to which they agree with the phrase "I want opioids" on a scale of 0 (Not-at-All) to 100 (Completely).
Time Frame: Averaged across the 8-week trial.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale (0-100)
Groups:
- Placebo: Maintenance on a daily dose of oral doxazosin (0 mg) for 4 weeks, Under placebo maintenance the effects of intranasal oxycodone were assessed.
- Doxazosin: Maintenance on a daily dose of oral doxazosin (16 mg, or the highest tolerated dose) for 4-weeks. Under doxazosin maintenance the effects of intranasal oxycodone were assessed.
Arm/Group | Placebo | Doxazosin
Number analyzed (Participants) | 2 | 2
units on a scale (0-100)
  Oxycodone 50 mg | 22.5 (12.6) | 27.3 (13.7)
  Oxycodone 0 mg | 33.6 (14.1) | 45.3 (15.1)
  Oxycodone 12.5 mg | 43.3 (14.9) | 50.6 (15.6)
  Oxycodone 25 mg | 30.5 (13.3) | 34.9 (13.7)
  Oxycodone 100 mg | 24.5 (11.4) | 26.1 (12.3)

ADVERSE EVENTS:
Time Frame: AEs and SAEs were assessed throughout the 8-week study period. Data are presented as a function of the 4-week period under which participants received placebo doxazosin, and the 4-week period during which they received active doxazosin.
Groups:
- Placebo Maintenance: Maintenance on a daily dose of oral doxazosin (0 mg) for 4 weeks.
- Doxazosin Maintenance: Maintenance on a daily dose of oral doxazosin (16 mg, or the highest tolerated dose) for 4-weeks.
Arm/Group | Placebo Maintenance | Doxazosin Maintenance
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 2/13 | 5/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Maintenance (N=13) | Doxazosin Maintenance (N=13)
Orthostasis (Cardiac disorders) | 2 (8) | 5 (13)
Bradychardia (Cardiac disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-12-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT03415581/Prot_000.pdf